CLINICAL TRIAL: NCT07325318
Title: Study on the Dose of Extracorporeal Shockwave Therapy for Treating Adhesive Capsulitis
Brief Title: Shockwave Dose for Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108-124-E
Record Dates: First submitted 2025-11-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Capsulitis, Shoulder
Keywords: Adhesive capsulitis; Range of motion; Extracorporeal shockwave therapy
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: two different shockwave doses are performed to treat adhesive capsulitis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extracoporeal sockwave therapy basic dose (Experimental): 3,000 pulses of shockwave per session as the basic treatment
  Interventions: Device: focused extracoporeal sockwave
- extracoporeal shockwave therapy high dose (Experimental): 6,000 pulses of shockwave per session as the high dose treatment
  Interventions: Device: focused extracoporeal sockwave

INTERVENTIONS:
Device: focused extracoporeal sockwave — Focused ESWT energy was initiated at level 5 (0.034 mJ/mm²) with a 4-Hz frequency and subsequently adjusted based on patient tolerance. After the application of coupling gel, different pulses were applied one fingerbreadth inferior to the anterior acromion, lateral to the acromion, and posterior to the acromion.

SUMMARY:
The investigators evaluated the therapeutic efficacy of different shockwave dosages for adhesive capsulitis and further examined the temporal effects and subgroup responses based on baseline range of motion

DETAILED DESCRIPTION:
The study compares two different shockwave treatment doses, each delivered as a single session to patients with adhesive capsulitis of the shoulder. We will measure shoulder range of motion before and after treatment and assess functional improvement using the Constant-Murley score. Finally, we will analyze changes in joint mobility at various post-treatment time intervals to evaluate the therapeutic effectiveness of the two shockwave dosing protocols.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥ 20 years
* first episode of adhesive capsulitis
* persistent shoulder pain with restricted motion for ≥ 3 months
* prior management limited to analgesic medications
* active abduction in the scapular plane ≤ 135°

Exclusion Criteria:

* shoulder or cervical pathology
* history of shoulder fracture, infection, or tumor
* previous shoulder surgery
* pacemaker presence
* pregnancy
* coagulopathy
* inability to complete follow-up assessments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
We assessed changes in shoulder range of motion using a standard goniometer before and after treatment with varying shockwave dosages | Before treatment, immediately after treatment, and at 1, 2, 4, 8, and 12 weeks post-treatment
  In patients receiving different doses of extracorporeal shockwave therapy for adhesive capsulitis, we assessed changes in shoulder range of motion before and after treatment using a standard goniometer. We will assess forward flexion, abduction, external rotation, and internal rotation. The better the range of motion, the better the treatment outcome.

SECONDARY OUTCOMES:
We assessed changes in shoulder functional outcomes using the Constant-Murley questionnaire before and after treatment with varying shockwave dosages | before treatment and 12 weeks posttreatment
  In patients receiving different doses of extracorporeal shockwave therapy for adhesive capsulitis, we evaluated changes in shoulder function by administering the Constant-Murley questionnaire both before and after treatment. The questionnaire includes four subcategories: pain score (maximum 15 points), activities of daily living (maximum 20 points), movement (maximum 40 points), and strength (maximum 25 points). The Constant-Murley Score has a maximum of 100 points, with higher scores indicating a better outcome."
The impact of changes over time before and after shockwave therapy on joint angle improvement | immediately after treatment and 1, 2, 4, 8, and 12 weeks posttreatment
  We analyzed the magnitude of joint angle changes at multiple time points to compare the therapeutic effects of the various shockwaves doses.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CJ, Huang CC, Yip HK, Yang YJ. Dosage effects of extracorporeal shockwave therapy in early hip necrosis. Int J Surg. 2016 Nov;35:179-186. doi: 10.1016/j.ijsu.2016.09.013. Epub 2016 Sep 21. PMID 27664561
- [Background] El Naggar TEDM, Maaty AIE, Mohamed AE. Effectiveness of radial extracorporeal shock-wave therapy versus ultrasound-guided low-dose intra-articular steroid injection in improving shoulder pain, function, and range of motion in diabetic patients with shoulder adhesive capsulitis. J Shoulder Elbow Surg. 2020 Jul;29(7):1300-1309. doi: 10.1016/j.jse.2020.03.005. PMID 32553435
- [Background] Gerdesmeyer L, Wagenpfeil S, Haake M, Maier M, Loew M, Wortler K, Lampe R, Seil R, Handle G, Gassel S, Rompe JD. Extracorporeal shock wave therapy for the treatment of chronic calcifying tendonitis of the rotator cuff: a randomized controlled trial. JAMA. 2003 Nov 19;290(19):2573-80. doi: 10.1001/jama.290.19.2573. PMID 14625334
- [Background] Yao G, Chen J, Duan Y, Chen X. Efficacy of Extracorporeal Shock Wave Therapy for Lateral Epicondylitis: A Systematic Review and Meta-Analysis. Biomed Res Int. 2020 Mar 18;2020:2064781. doi: 10.1155/2020/2064781. eCollection 2020. PMID 32309425
- [Background] Walker-Bone K, Palmer KT, Reading I, Coggon D, Cooper C. Prevalence and impact of musculoskeletal disorders of the upper limb in the general population. Arthritis Rheum. 2004 Aug 15;51(4):642-51. doi: 10.1002/art.20535. PMID 15334439
- See also: The website describes the shockwave device used in the study as well as the underlying treatment principles. — https://www.richard-wolf.com/en/disciplines/shockwaves/piezowave2